CLINICAL TRIAL: NCT04883281
Title: DARTBOARD: a Prospective Randomized Phase II Study of Daily Adaptive Radiotherapy to Better Organ-at-Risk Doses in Head and Neck Cancer
Brief Title: A Prospective Study of Daily Adaptive Radiotherapy to Better Organ-at-Risk Doses in Head and Neck Cancer
Acronym: DARTBOARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Sher, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0401
Record Dates: First submitted 2021-04-27; First posted 2021-05-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Involved Nodal Radiotherapy with conventional margins w or w/o chemotherapy (Active Comparator): If a patient loses a significant amount of weight on treatment, or the tumor contour changes substantially, repeat CT simulation and re-planning is allowed in the CM arm. However, the gross tumor volume may not be reduced due to tumor shrinkage. The original extent of disease must be included in the replanned GTV.
  Interventions: Radiation: Intensity modulated radiation therapy (IMRT) with or without chemotherapy; Drug: cisplatin, cetuximab, or carboplatin-paclitaxel
- Involved Nodal Radiotherapy with marginless Daily Adaptive Radiotherapy w or w/o chemotherapy (Experimental): Patients in the ML/DART Arm will have their radiation plan adapted with every fraction. The adaptation process will be performed automatically on the Varian Ethos adaptive therapy software under the supervision of the treating physician.
  Interventions: Radiation: Intensity modulated radiation therapy (IMRT) with or without chemotherapy; Drug: cisplatin, cetuximab, or carboplatin-paclitaxel

INTERVENTIONS:
Radiation: Intensity modulated radiation therapy (IMRT) with or without chemotherapy — Intensity modulated radiation therapy (IMRT) with or without chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel)
Drug: cisplatin, cetuximab, or carboplatin-paclitaxel — chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel)

SUMMARY:
Varian Medical Systems has recently deployed a completely novel radiation treatment system called EthosTM, a first-of-its-kind system that allows for daily adapative radiotherapy (DART), such that the treatment for that day can be created on-the-fly based on the patient's current positioning and anatomy. This system is commercially-available and FDA-approved, and UTSW Radiation Oncology has installed two such units. The ability to adjust the dose delivery every day means both that adaptive therapy is possible with every fraction and that the PTV margin can be dramatically reduced/eliminated, since investigators are treating for that day's patient setup. Investigators are therefore proposing a randomized trial using DART with near marginless (ML) setup margins (a 1 mm margin will be retained for intrafractional motion).

DETAILED DESCRIPTION:
IMRT with daily cone-beam computed tomography (CBCT) set up is the current recommended radiation technique for head and neck squamous cell carcinoma. The conformality of IMRT has made it possible to reduce dose to normal tissues, but it also predisposes the treatments to drastic delivered dose deviations due to changes in the patient (e.g. weight loss, muscle atrophy, or normal tissue edema) or in the tumor (e.g. treatment response or treatment related edema). These changes can create poor coverage and/or cold spots in the tumor and increased coverage and/or hot spots in the normal organs at risk. Image guidance with CBCTs can help reduce set up error between treatments, but image guidance can't adjust for these patient or tumor changes.

Adaptive radiotherapy (ART) is the process of replanning the patient's radiation plan by adjusting the target structures, organs at risk structures, and optimal radiation delivery during the radiation therapy course. ART allows treating physicians to account for all the patient or tumor changes that can't be currently resolved with image guidance. Previously, ART was a prohibitively resource and time-consuming process that could only be performed once or twice during a conventional 6.5 to 7-week head and neck radiation treatment course in select patients with substantial structural changes. However, with the recent advent of adaptive software, ART can now be performed on a daily basis.

The data on the possible advantages of ART in head and neck cancer is still limited to small, mostly pre-clinical studies. In a feasibility study, five patients with locally advanced HPV-positive oropharynx cancer undergoing definitive chemoradiation underwent an MRI every two weeks during their treatment. The results showed an average decrease in the primary tumor GTV volume of 44%, 90%, and 100% and an average decrease in the nodal GTV volume of 25%, 60%, and 80% by at weeks 2, 4, and 6 weeks, respectively. Another similar study on eight patients saw an average 70% GTV volume reduction by week 6.

In addition to tumor coverage, parotid glands are of particular interest in ART because of their radiosensitivity and association with xerostomia and decreased quality of life. Toxicity of salivary glands are related to dose as a continuous variable, so even modest decreases in dose can have a clinical impact. The average volume of the parotids has been reported to decrease as much as 14.7%, 37%, and 48% by the end of weeks 2, 4, and 7. The parotid glands also appear to shift superiorly and medially during treatment. Feasibility ART studies have shown that the dose to the parotid may decrease by as much as 5.5 Gy with ART. Therefore ART holds the promise of preserving the expected dose distribution to salivary OARs, improving long-term patient outcomes.

The ability to ensure coverage of the target structures and proper avoidance of organs at risk on a daily basis also greatly improves the confidence of the daily set-up and targeting. Current recommended radial PTV margins with daily CBCT are 3-5 mm, with even larger margins recommended for patients at risk of larger inter-fraction variability. These PTV margins are built to ensure the disease is not missed by the treatment due to daily setup error. However, these margins also significantly increase the irradiated volume, since the volume increases exponentially with each additional millimeter. Therefore, decreasing margins, even by a few millimeters, can results in large changes in treatment volume and improvement in toxicity.

In a retrospective Danish analysis of patients treated with 5 mm versus 3 mm PTV margins, Navran et al. noted that acute grade 3 toxicity (65% vs 53.8%, p = 0.008) and late grade 3 dysphagia (20.4% vs 11.1%, p = 0.012) were significantly lower in the smaller margin group. There were no differences in disease outcomes between the two groups. In a retrospective study analyzing the benefit of changing the margin on gross disease from 8 mm to 5 mm, just a 3 mm difference, Samuels et al. found that plans with the smaller PTV margin had a clinically meaningful improvement in the normal tissue complication probability for the ipsilateral parotid gland and contralateral submandibular gland when compared to conventional PTV margin plans. In fact, 40% of patients would have theoretically experienced an improvement in the function of both of these glands, just by modestly shrinking the PTV.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-proven diagnosis of squamous cell carcinoma of the oropharynx, larynx, or hypopharynx. Squamous cell carcinoma of unknown primary is not allowed.
* Patients must have clinically or radiographically evident measureable disease at the primary site and/or nodal stations. Diagnostic lymph node excision (< 2 nodes) is also allowable.
* Patients may undergo a diagnostic or therapeutic transoral resection for a T1-2 tonsil or base of tongue cancer.
* Clinical stage I-IVB (AJCC, 7th edition); stages I-II glottic cancer are excluded
* Age ≥ 18 years.
* ECOG Performance Status 0-2
* Negative serum or urine pregnancy test within 2 weeks before registration for women of childbearing potential.
* Neck CT and/or neck MRI, and PET-CT (at least skull-to-thigh).
* Ability to understand and the willingness to sign a written informed consent.
* All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* Distant metastasis.
* Inability to undergo PET-CT.
* Stage I and II glottic carcinoma.
* Gross total excision of both the primary and nodal disease.
* Synchronous non-skin cancer primaries outside of the oropharynx, larynx, and hypopharynx except for low- and intermediate-risk prostate cancer and synchronous well-differentiated thyroid cancer; in the latter case, surgery may occur before or after treatment, provided all other eligibility criteria are met.
* Prior invasive malignancy with an expected disease-free interval of less than 3 years.
* Prior systemic chemotherapy for the study cancer; prior chemotherapy for a remote cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields.
* Subjects may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the chemotherapy agents in this study (if necessary).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
* pregnant or nursing women
* History of severe immunosuppression, including HIV, and organ or autologous or allogeneic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Xerostomia Questionnaire (XQ) | 1 year
  1-year score on the Xerostomia Questionnaire (XQ) to determine the difference in chronic xerostomia between patients treated with conventional INRT versus ML DART INRT. The XQ score at one year will be compared between the arms using a two-sided t test.

SECONDARY OUTCOMES:
Development of acute and chronic toxicity in patients treated with and without DART | 1 year
  Incidence of acute grade 2+ radiation dermatitis, acute and chronic grade 3+ dysphagia, acute grade 3+ mucositis, and chronic grade 2+ soft tissue and osteonecrosis. Each toxicity endpoint will be compared between the arms using a Fisher exact test.
Risk of locoregional recurrence with and without DART | 1 year
  Cumulative incidence of locoregional recurrence, as confirmed by biopsy. The cumulative incidence of locoregional and distant failure will be estimated using cumulative incidence statistics, with death serving as the competing risk. The two arms will be compared using Gray's test.
Patient reported outcomes | 1 year
  Patient Reported Outcomes (PRO): EORTC QLQ-30 Global Score, EORTC HN 35 Pain and Senses Scores, MDADI Composite Score Each of the patient reported outcomes are single numeric scores that are collected at baseline, 1, 3, 6, and 12 months from treatment. Patients with disease recurrence will be excluded. At each individual time point, the differences between the arms in the changes of these outcomes between baseline to that timepoint will be compared using a t-test and analyzed longitudinally using generalized estimated equations (GEE).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sher DJ, Avkshtol V, Lin MH, Wang J, Chen L, Liao CY, Hughes R, Domal S, Ahn C, Moon DH. Impact of daily adaptive head and neck radiotherapy on toxicity and quality of life: results of the DARTBOARD phase II randomized trial. J Natl Cancer Inst. 2025 Dec 1;117(12):2488-2494. doi: 10.1093/jnci/djaf232. PMID 40833933